CLINICAL TRIAL: NCT01156454
Title: Specimen X-Rays of Removed Axillary Lymph Nodes to Guide Pathological Sampling (GPS)
Brief Title: Specimen X-Rays of Removed Axillary Lymph Nodes to Guide Pathological Sampling
Acronym: GPS
Status: Completed | Type: Observational
Sponsor: University of Arkansas (Other)
Collaborators: Tenenbaum Family Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 111743
Record Dates: First submitted 2010-06-24; First posted 2010-07-02 (Estimated); Last update posted 2016-12-23 (Estimated); Status verified 2016-12

CONDITIONS: Breast Cancer
Keywords: sentinel lymph node dissection; radiology; X-ray identification of nodes in a surgical specimen
MeSH Terms: conditions — Breast Neoplasms | interventions — X-Rays

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Surgery followed by x-ray assessment: After nodes are removed they are taken to radiology to be x-rayed
  Interventions: Procedure: X-ray

INTERVENTIONS:
Procedure: X-ray — surgical specimen taken to radiology and contents x-rayed

SUMMARY:
X-ray mapping of sentinel lymph nodes and/or axillary tissue will assist pathologists in their ability to identify the number and location of lymph nodes as well as more accurately section lymph nodes contained in surgical specimens.

ELIGIBILITY:
Inclusion Criteria:

Males or females of all races and ethnicities

* ≥ 18 years of age
* Must be scheduled for breast cancer surgery which includes a sentinel lymph node biopsy and/or axillary dissection

Exclusion Criteria:

• Any person whose final pathology could be compromised in any way by the X-ray procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Males or females of all races and ethnicities, must be equal to or greater than 18 years of age, scheduled for breast cancer surgery that includes sentinel node biopsy and/or axillary dissection
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2009-11; Primary Completion 2011-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Identification of lymph nodes | Within the first 30 minutes after specimen is removed from the body
  To determine if plain x-ray films obtained from the sentinel node/axillary dissection specimen can facilitate the identification of the lymph nodes and increase the average number of lymph nodes recovered by the pathologist.
Identification of affected area in node | Within the first 30 minutes after specimen is removed from the body
  To determine whether plain x-ray films obtained from the sentinel node/axillary dissection specimen can help direct the pathologist to the correct part of the node (the portion containing disease) to sample.

CONTACTS AND LOCATIONS:
Overall Officials: V. Suzanne Klimberg, MD, Principal Investigator — UAMS
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

REFERENCES:
- [Result] Johnson CB, Korourian S, Badgwell BD, Fincher RL, Dell CM, Don Bice C, Boneti C, Westbrook KC, Klimberg VS. Sensitivity of axillary specimen x-ray to predict nodal count and positivity. Ann Surg Oncol. 2011 Oct;18(11):3181-6. doi: 10.1245/s10434-011-1959-x. Epub 2011 Aug 23. PMID 21861231